CLINICAL TRIAL: NCT03640507
Title: The Effect of Vaginal Preparation With Chlorhexidine-alcohol vs. Povidine-iodine vs. Saline on Vaginal Bacteria Colony Counts in Pregnant Women
Brief Title: Vaginal Preparation With Chlorhexidine-alcohol vs. Povidine-iodine vs. Saline
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Yiping Weng Han, Professor of Microbial Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: AAAR4891
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-05

CONDITIONS: Cesarean Section; Infection; Surgical Site Infection
Keywords: vaginal preparation; antisepsis; C-section
MeSH Terms: conditions — Infections; Surgical Wound Infection | interventions — Chlorhexidine; Ethanol; Povidone-Iodine; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chlorhexidine-alcohol (Active Comparator): Subjects will receive vaginal preparation with chlorhexidine-alcohol.
  Interventions: Drug: Chlorhexidine-alcohol
- Povidine-iodine (Active Comparator): Subjects will receive vaginal preparation with povidine-iodine.
  Interventions: Drug: Povidine-iodine
- Saline (Placebo Comparator): Subjects will receive vaginal preparation with sterile saline.
  Interventions: Drug: Sterile saline

INTERVENTIONS:
Drug: Chlorhexidine-alcohol — Intervention is a 30-second vaginal preparation or topical wash with three chlorhexidine-alcohol 0.5% solution-soaked sponge sticks.
  Other Names: Chlorohexidine Gluconate (CHG)
  Arms: Chlorhexidine-alcohol
Drug: Povidine-iodine — Intervention is a 30-second vaginal preparation or topical wash with three povidine-iodine 10% solution-soaked sponge sticks.
  Other Names: Betadine
  Arms: Povidine-iodine
Drug: Sterile saline — Intervention is a 30-second vaginal preparation or topical wash with three sterile saline-soaked sponge sticks.
  Other Names: Sodium chloride 0.9%
  Arms: Saline

SUMMARY:
The purpose of this study is to see whether chlorhexidine is superior to povidine-iodine vaginal antisepsis at reducing bacteria colony counts in pregnant women by comparing three groups: vaginal washing with chlorhexidine-alcohol, vaginal washing with povidine-iodine, and vaginal washing with saline alone.

DETAILED DESCRIPTION:
This is a prospective trial of vaginal preparation (or vaginal cleansing/washing) on late preterm and term pregnancies admitted to Labor & Delivery unit for cesarean delivery with three arms. Randomization allocation would be performed in 1:1:1 fashion for vaginal preparation with chlorhexidine-alcohol, povidine-iodine, and saline washes. A saline wash group is included to determine if the act of cleansing the vagina with a sponge alone reduces bacterial colony counts.

ELIGIBILITY:
Intervention Group (vaginal preparation)

Inclusion Criteria:

* Pregnant women admitted for cesarean delivery
* Gestational age greater than or equal to 34 weeks

Exclusion Criteria:

* Rupture of membranes or active labor
* Chorioamnionitis (prior to enrollment)
* Recent (within 4 weeks) antibiotic exposure
* Maternal HIV infection or immunocompromised state
* Known allergy to shellfish, iodine, or chlorhexidine

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yiping Han, PhD, Principal Investigator — Columbia University Department of Microbiology and Immunology
Locations (1):
- New York Presbyterian Hospital at Columbia University and Children's Hospital of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duffy CR, Garcia-So J, Ajemian B, Gyamfi-Bannerman C, Han YW. A randomized trial of the bactericidal effects of chlorhexidine vs povidone-iodine vaginal preparation. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100114. doi: 10.1016/j.ajogmf.2020.100114. Epub 2020 Apr 15. PMID 33345865
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be recruited in-person only by study investigators/trained research personnel after admission to labor and delivery prior to administration of sedatives, anesthetics, or other mental-altering medications (note: some patients included in study will be in labor and may have already received regional anesthesia).
Pre-assignment Details: Participants need to be confirmed to be undergoing a Cesarean procedure.
Period: Overall Study
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline
Started | 10 | 9 | 11
Completed | 10 | 9 | 10
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline | Total
Number analyzed (Participants) | 10 | 9 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (5.8) | 34.3 (4.9) | 37.8 (4.6) | 35.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 10 | 29
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 11
  Not Hispanic or Latino | 6 | 5 | 7 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 6 | 8 | 23
  Black | 0 | 0 | 1 | 1
  Other | 1 | 3 | 1 | 5
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.0 (7.5) | 32.0 (5.5) | 35.6 (9.4) | 33.6 (7.6)
Insurance Payer [Count of Participants; unit: Participants]
  Private | 7 | 8 | 8 | 23
  Public | 3 | 1 | 2 | 6
Parity [Median (Inter-Quartile Range); unit: prior deliveries] | 1 [0 to 1] | 1 [1 to 1] | 1 [0 to 1] | 1 [0 to 1]
GBS positivity [Count of Participants; unit: Participants] — As assessed by routine late third trimester screening (i.e. rectovaginal culture).
  Participants | 3 | 2 | 4 | 9
Co-morbidity [Count of Participants; unit: Participants] — Includes maternal cardiac disease, diabetes on medications, hypertensive disease and cholestasis of pregnancy
  Participants | 2 | 3 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Post-intervention Aerobic Bacterial Colony Counts
Description: Vaginal cultures are collected after the vaginal preparation intervention. These undergo serial dilutions and are incubated on Tryptic Soy Agar for seven days. Bacteria colony counts were determined by blinded investigators on day 7.
Time Frame: From intervention to 7 days post
Measure: Mean (Standard Error); unit: Log (CFU/mL)
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline
Number analyzed (Participants) | 10 | 9 | 10
Log (CFU/mL) | 2.959 (0.624) | 0.945 (0.438) | 5.104 (0.299)

2. Primary Outcome: Post-intervention Anaerobic Bacterial Colony Counts
Description: as for outcome 1
Time Frame: From intervention to 7 days post
Measure: Mean (Standard Error); unit: Log (CFU/mL)
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline
Number analyzed (Participants) | 10 | 9 | 10
Log (CFU/mL) | 4.934 (0.514) | 2.637 (0.682) | 5.804 (0.212)

3. Secondary Outcome: Baseline Aerobic Bacterial Colony Counts
Description: Vaginal cultures are collected immediately prior to the vaginal preparation intervention. These undergo serial dilutions and are incubated on Tryptic Soy Agar for seven days. Bacteria colony counts were determined by blinded investigators on day 7.
Time Frame: From intervention to 7 days post
Measure: Mean (Standard Error); unit: Log (CFU/mL)
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline
Number analyzed (Participants) | 10 | 9 | 10
Log (CFU/mL) | 5.942 (0.538) | 5.667 (0.437) | 6.480 (0.330)

4. Secondary Outcome: Baseline Anaerobic Bacterial Colony Counts
Description: as for outcome 3
Time Frame: From intervention to 7 days post
Measure: Mean (Standard Error); unit: Log (CFU/mL)
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline
Number analyzed (Participants) | 10 | 9 | 10
Log (CFU/mL) | 7.096 (0.240) | 6.745 (0.339) | 7.145 (0.316)

5. Other Pre Specified Outcome: Number of Participants Diagnosed With Postpartum Infections.
Description: Chart review to assess any maternal infections diagnosed during postpartum hospitalization or at the time of the postpartum visit.
Time Frame: Up to six weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline
Number analyzed (Participants) | 10 | 9 | 10
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to 6 weeks postpartum
Arm/Group | Chlorhexidine-alcohol | Povidine-iodine | Saline
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/11

LIMITATIONS AND CAVEATS:
Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03640507/Prot_SAP_000.pdf